CLINICAL TRIAL: NCT07270276
Title: The Impact of Dry Needling on Electrophysiological and Ultrasound-based Biomarkers for Myofascial Pain
Acronym: ENCOMPASS-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Seward Rutkove, Department of Neurology Chair, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P000944; R33AT012284 (NIH)
Record Dates: First submitted 2025-11-19; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Trigger Point in Trapezius Muscle
Keywords: Myofascial Pain; Trigger Point; Myofascial Pain Syndrome; Trapezius Muscle Pain
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dry Needling Treatment Group (Experimental)
  Interventions: Procedure: Dry Needling
- Sham/Placebo Treatment Group (Placebo Comparator)
  Interventions: Procedure: Sham Treatment

INTERVENTIONS:
Procedure: Dry Needling — A physical therapy and pain management technique where a small is inserted into a trigger point (tight, tender spots in the muscle that cause pain) and maneuvered to provide pain relief.
  Arms: Dry Needling Treatment Group
Procedure: Sham Treatment — Treatment where a sham treatment will be administered which does not directly target the trigger point. Subjects will not be able to tell the difference between dry needling and sham treatment.
  Arms: Sham/Placebo Treatment Group

SUMMARY:
The goal of this interventional study is to determine how well dry-needling can treat pain in people with Myofascial Pain Syndrome. The main questions it aims to answer are:

* Does dry needling improve pain for people with a trigger point (a tender, tight spot in the muscle)?
* How well can Electrical Impedence Myography (EIM), Myofiber Threshold Tracking (TT), and Ultrasound (US) detect changes in the muscle related to dry needling treatment?

Researchers will compare dry needling to a placebo (a treatment that does not enter the trigger point) to see if dry needling works to treat Myofascial Pain Syndrome with trigger points in the trapezius muscle (the muscle that extends over the back of the neck and shoulders), as measured by these three outcome measures (EIM, US, TT).

Participants will:

* Visit the clinic twice: once to receive dry needling treatment, and once for a follow-up
* Have muscle measurements taken before treatment and at follow-up
* Have a daily survey to record the intensity of their pain

DETAILED DESCRIPTION:
Pre-Screening:

Participants will be pre-screened to assess eligibility. The questionnaire can be completed on the phone, online in a survey, or in person. Medical records will also be reviewed. Eligible participants will schedule an on-site visit.

Study Visit #1:

In most cases the following sessions will occur on one day, unless due to scheduling conflicts separate sessions must be scheduled.

1. Eligibility & Screening: Baseline review of medical history and medication will be done to ensure eligibility. Informed consent will be taken from participants. Demographic data will be taken. This will take approximately one hour.

   The following baseline procedures will occur:
2. Trigger point will be identified in the trapezius muscle, and marked with a marker by a physician.
3. Electrical Impedance Myography (EIM) - a trained technician will apply several small sticky pads (electrodes) to different parts of the subject's muscle and a very tiny electrical current will be applied that they will not feel. Several measurements will be done their muscle. This will take approximately 10 minutes
4. Ultrasound (US) - a trained technician will apply a small amount of gel to the skin. They will hold a small hand-held device on the skin and will measure the muscle. The gel is easily cleaned off of the skin when the testing is complete. This will take approximately 20 minutes.
5. Threshold Tracking (TT) - TT tests how quickly muscle responds to stimulation. The muscle is stimulated using a small needle which is placed superficially in their trapezius muscle. The subject will feel a small needle prick which should be less uncomfortable than having blood drawn. Electrodes (small sticky pads) are placed a short distance from the needle over the muscle. When their muscle is stimulated with the needle, the time it takes for the muscle to react is measured by the electrodes. This procedure will last 30 minutes and creates a tingling feeling.
6. Algometry - a controlled pressure will be applied to the trigger point to measure pain response. This will take 5 minutes.
7. Questionnaires- Subjects will be asked to complete some brief questionnaires about their pain, mood, and sleep.
8. Dry needling treatment or sham procedure will be administered by a physician. This will take 5-10 minutes.

Home Period:

1. Subjects will be asked to re-apply the marker spot made at their first visit as it fades. This is so investigators can use the same spot for testing at the next visit.
2. A pain survey will be taken daily either online, by phone, or on paper.

Study Visit #2:

This visit will occur approximately two weeks after the intervention. It will take around 2 hours.

1. Imaging and testing measures including EIM, TT, US, and algometry will be performed.
2. Questionnaires taken at baseline, and two additional ones, will be administered.
3. Adverse events and pain medication regimens will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-80
* Presence of active trigger points with involvement of upper trapezius
* Able to manage breakthrough pain with acetaminophen only, excluding stable doses of pain medications at time of enrollment, which can be continued

Exclusion Criteria:

* Multiple active trigger points in the trapezius muscle if physician assessment concludes that this may interfere with subject's ability to detect changes in pain improvement from trigger point therapy
* Presence of cervical radicular pain, superimposed neuromuscular disease or condition that, in the opinion of the investigator, could confound interpretation of the data acquired from trapezius.
* Fibromyalgia or other generalized pain condition
* Opioid usage in the past 3 months
* Active substance use disorder
* Not on a stable dose for at least two weeks prior to study enrollment or unwilling to maintain a stable dose for duration of the study of the following drugs:

  1. SSRIs, such as citalopram, escitalopram, fluoxetine, sertraline,
  2. SNRIs, such as duloxetine, milnacipran, and venlafaxine
  3. Tricyclic antidepressants, such as notritptyline, amitriptyline, and desipramine
  4. Alpha 2 delta ligands: pregabalin, gabapentin
  5. Specific anti-epileptics: topiramate, lamotrigine, oxcarbazepine, and phenytoin
  6. Other: quinidine, mexiletine, and dalfampridine
* Skin allergy or sensitivity that would preclude the use of adhesive electrodes
* Significant systemic or psychiatric illness that in the opinion of the site Investigator would interfere with the individual's ability to participate in the trial
* Anticoagulation (with coumadin, clopidogrel, or direct oral anticoagulants; aspirin acceptable)
* TrP needle-based therapy in the past six weeks of the TrP to be studied
* Body mass index > 35 kg/m2
* Other factor that in the opinion of the site investigator would interfere with the ability to perform the study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Excitability threshold tracking (TT) | From enrollment to end of treatment follow up (2 weeks)
  The secondary outcome will be maximum latency change with a conditioning stimulus

SECONDARY OUTCOMES:
Muscle ultrasound | From enrollment to end of treatment follow up (approximately 2 weeks)
  Echointensity
Electrical Impedance Myography (EIM) | From enrollment to end of treatment follow up (2 weeks)
  The primary outcome will be 100 kHz phase angle in EIM
Algometer Measurement Device Output | From enrollment to end of treatment follow up (2 weeks)
  The algometer is a simple pressure measurement tool which is placed directly over the trigger point. The examiner pushes down on the algometer, gradually increasing the pressure applied. The participant than verbally tells the examiner when they feel pain; the procedure is then terminated, and the examiner records the algometer pressure (measured in kg/cm^2) at the instant of pain as the result. A lower value indicates greater pain sensitivity.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
A final, complete, cleaned, and coded study data set will be provided for public access including the appropriate data dictionaries and case report forms on the Vivli data repository platform.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD will be available following completion of all planned analyses and manuscripts.
Access Criteria: We will make the data and associated documentation available to a NIH HEAL Initiative approved Central Data Repository, such as Vivli.